CLINICAL TRIAL: NCT00907660
Title: A Randomized Trial Comparing Two Doses of Portion-Controlled Foods Within a Primary Care Weight Loss Program
Acronym: PCPCWLS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-0054; K24DK065018 (NIH)
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; Meal replacements; Health services research
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Nutrition Assessment; Behavior Therapy; Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full Dose (Active Comparator): Provision of 8 weight loss counseling sessions, calorie guide, pedometer, meal plan, and 2 meals per day of portion-controlled foods (shakes and entrees)
  Interventions: Behavioral: Weight loss counseling; Dietary Supplement: Portion-Controlled Foods
- Half dose (Experimental): Provision of 8 weight loss counseling sessions, calorie guide, pedometer, meal plan, and 1 meal per day of portion-controlled foods (shakes and entrees)
  Interventions: Behavioral: Weight loss counseling; Dietary Supplement: Portion-Controlled Foods

INTERVENTIONS:
Behavioral: Weight loss counseling — Monitoring of weight; review of food and physical activity records; counseling to reduce calorie intake by 500-1000 calories per day
  Other Names: Dietary counseling; Behavior modification; Diet and exercise
Dietary Supplement: Portion-Controlled Foods — Consumption of shakes, meal bars, and prepared entrees for 2 out of 3 meals per day during the 14 weeks of the study. "Full dose" patients are provided with both meals by the study; "half dose" patients are provided with one out of two meals by the study.
  Other Names: Meal replacements

SUMMARY:
We hypothesize that individuals provided with 1 meal per day of portion-controlled foods (shakes and prepared entrees) will lose as much weight as individuals provided with 2 meals per day of portion-controlled foods. The study is designed to assess whether equal weight loss can be achieved at a lower cost to the health care system (or health care payer), with patients contributing some of the cost of their own treatment.

DETAILED DESCRIPTION:
The study has two goals. First, it will assess the efficacy of a weight loss program, using a combination of counseling by peer weight coaches and portion-controlled foods. Second, the study will test the effect of varying the "dose" of portion-controlled foods provided to patients by randomly assigning individuals to receive half or all of the food required to follow a meal replacement regimen. The primary endpoint of the study will be weight change. Secondary endpoints will include adherence to the recommended eating plan, health-related quality of life, as well as changes in waist circumference and blood pressure. The provision of "half-dose" portion-controlled foods (1 meal per day) is hypothesized to be non-inferior to provision of "full-dose" (2 meals per day). The goal of non-inferiority is important because it can demonstrate that health care payers wishing to support weight loss programs can achieve equivalent results at a lower cost. All patients have the choice regarding their use of portion-controlled foods in the study, and no patients will be asked to leave the study because of non-adherence.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the University Medicine Denver, University Medicine Anschutz, and A.F. Williams clinics meeting the following criteria
* Age 18 or older
* Able to keep a food record for 3 days prior to study entry
* Able to give informed consent
* Willing to accept randomization to either treatment condition, to attend all sessions, and to complete study-related assessments
* Body mass index (BMI) ≥ 30 kg/m2 and < 50 kg/m2
* Elevated waist circumference (≥ 88 cm for women, ≥ 102 cm for men) + any one of the following:
* Glucose intolerance (fasting glucose ≥ 100 or non-fasting glucose ≥ 140, including type 2 diabetes); individuals taking medications for diabetes qualify automatically
* Elevated blood pressure (≥130/85), including hypertension (≥140/90); individuals taking anti-hypertensive medication qualify automatically
* Hypertriglyceridemia (TG ≥ 150); individuals taking lipid-lowering medications qualify automatically
* Decreased high-density lipoprotein (HDL) cholesterol (< 40 for men, < 50 for women)
* Obstructive sleep apnea

Exclusion Criteria:

* Medical conditions in which significant weight loss is normally contraindicated (e.g. pregnancy, congestive heart failure requiring diuretics, poorly controlled diabetes, Stage 4 or 5 chronic kidney disease, clinically evident cirrhosis, other severe internal organ disease); exceptions may be made if a referring physician documents that it is safe and appropriate for the individual to lose weight
* Treated for cancer within the past 5 years, except for basal cell or squamous cell skin cancer; exceptions may be made with written permission from a physician
* Weight gain or loss of ≥5% of weight in the past 6 months; patients who have not been weight stable may be re-screened in 3 months
* Concurrent use of corticosteroids or second-generation antipsychotic medications (exceptions may be made for individuals using these medications who have been weight stable for 6 months)
* Psychiatric diagnoses likely to affect adherence to a research study protocol (e.g., poorly controlled schizophrenia, active substance abuse)
* Prior or planned bariatric surgery
* Participation in an organized weight loss program (e.g., Weight Watchers) at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Weight change | 14 weeks

SECONDARY OUTCOMES:
Health-related quality of life | 14 weeks
Blood pressure | 14 weeks
Waist circumference | 14 weeks
Body mass index | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adam G Tsai, MD, MSCE, Principal Investigator — University of Colorado, Denver
Locations (1):
- Center for Human Nutrition, Denver, Colorado, United States